CLINICAL TRIAL: NCT00200980
Title: Importance of Non-Acid Reflux in Moderate and Severe Asthma
Brief Title: Importance of Non-Acid Reflux in Asthma in Children
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry)
Other Study IDs: 0504609
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Asthma; Gastroesophageal Reflux
MeSH Terms: conditions — Asthma; Gastroesophageal Reflux

SUMMARY:
The purpose of the study is to follow the medical course of children with moderate to severe asthma and see how this relates to whether they have acid of non-acid gastroesophageal reflux

DETAILED DESCRIPTION:
Research Plan

Hypothesis and Specific Aims:

Asthma and gastroesophageal reflux are both common medical conditions in infants and children as in adults, and often co-exist (Gibson 2002, Andze, 1991). Though an association with overt reflux disease and asthma is well described and accepted, occult acid reflux has also been shown to be associated with asthma. The vexing question has been whether non-acidic reflux exacerbates asthma, particularly moderate to severe asthma. Current approaches and the extensive literature to date have dealt with the role of acid reflux only, and hence medical management is dominated by gastric acid suppression strategies recently outlined by a consensus statement from the North American Society of Pediatric Gastroenterology, Hepatology and Nutrition (Rudolph 2001). Based on this consensus, and randomized double blind studies in adults, our strategy is to now use long-term proton pump inhibitors. Clinically, this intervention has limited impact, and treatment failures are common. Now that non-acid gastroesophageal reflux can be measured with the combined impedance and pH probe, the role of non acid reflux can finally be evaluated. Our experience thus far confirms findings of limited published pediatric studies using a significant role for non-acid reflux in these "non -responders", and indeed suggests a greater role of non-acid GER in extra-esophageal disorders in general. This new tool supercedes the standard pH probe. Currently the standard of care for moderate to severe asthma is evaluation for association with gastroesophageal reflux. These cases at NCC-Wilmington undergo 24 hour combined impedance and pH study. With the advent of this new tool at NCC-Orlando also, we plan to combine resources at several sites to accumulate data on prevalence of acid and non-acid reflux in asthma. This would be an effective use of data retrieval attributes of EPIC. Future studies looking at the impact of type of refluxate on bronchospasm, parenchymal damage, and even chronic pulmonary vascularity changes prospectively would then be set up. Since currently we have no specific recommendations for medical treatment of non-acid GER, therapeutic strategies, either with existing or newer motility agents, could also be evaluated in the future to develop practice guidelines.

Specific Aim:. What is the prevalence of acid and non-acid GER in moderate to severe asthma patients referred for GI evaluation

Prevalence of acid and non-acid gastroesophageal reflux in children 1 to 18 yrs with moderate asthma and severe asthma, referred for evaluation of gastroesophageal reflux at NCC-Wilmington, New Jersey, and NCC-Orlando will be obtained. This information will be extracted from EPIC templates that have current standards of care incorporated.

ELIGIBILITY:
Inclusion Criteria:

Moderate to Severe Asthma in Children 1 - 18 years

Exclusion Criteria:

Antireflux surgery Unable to have 24 hr reflux study completed

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Devendra I Mehta, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Nemours Children's Clinic, Orlando, Florida, United States